CLINICAL TRIAL: NCT04117282
Title: Effect of Antigravity Shoes on Improving the Quality of Gait in Children With Spastic Diplegia (Using 2 D Gait Analysis)
Brief Title: Effect of Antigravity Shoes on Improving the Quality of Gait in Children With Spastic Diplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nahla Mohamed Ibrahim, Doctoral degree (lecturer), Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pediatric physical therapy
Record Dates: First submitted 2019-10-02; First posted 2019-10-07 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: 2 groups study and control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): 15 children received the regular exercise program including classical gait training for diplegic children (30 minutes exercises + 30 minutes gait training)
  Interventions: Other: gait training
- study group (Experimental): 15 diplegic child received the same exercise program including the use of the antigravity shoes for gait training (30 minutes exercises + 30 minutes gait training)
  Interventions: Other: gait training

INTERVENTIONS:
Other: gait training — training for improving the quality of gait through adjusting gait cycle phases time and improving the functional level and independence during gait
  Other Names: gait rehabilitation

SUMMARY:
Improving the quality of gait in the diplegic children is a major concern in the rehabilitation program. Thirty children with spastic diplegia were distributed equally into 2 groups, group A (control) and group B (study). Group A had received the traditional physical therapy program for 30 minutes and 30 minutes traditional gait training, while group B had received 30 minutes gait training with antigravity shoes in addition to the traditional exercise program for 30 minutes, percentage of stance and swing phase of gait were measured by 2 D gait analysis for children of both groups pre and after 3 successive months of treatment program, also function level of gait were assessed pre and post treatment by GMFCS .

DETAILED DESCRIPTION:
Thirty children with spastic diplegia, their age ranged from 6 to 8 years old, were distributed equally into 2 groups: group A (control) and group B (study) They could walk with limitation or holding on according to GMFCS (level II &III). (Palisano et al., 2008). Increased time for stance phase and decreased swing phase time was recorded when evaluated by 2D gait analysis.

Control group (A):

The children in this group had received traditional physical therapy exercise program designed for those cases for 30 minutes in addition to gait training program for 30 minutes / day, 3 times / week for 3 successive months.

Study group (B):

The children in this group received the same traditional exercise program for 30 minutes in addition to gait training program for 30 minutes using the antigravity shoes.

evaluation was done before and after treatment. treatment include traditional exercises for gait and balance for both groups in addition to use the antigravity shoes for study group.

ELIGIBILITY:
Inclusion Criteria:

* 30 diplegic children of both gender aged from 6 to 8,
* GMFCS levelII and II . has gait defecits including percentage of gait cycles.

Exclusion Criteria:

* recent surgical intervention.
* orthopedic deformity in lower limbs.
* sever vision or hearing problems.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-02-03 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
gait time percentage for right lower limb | after 3 months of treatment
  the time of stance and swing phases as a percentage for right lower limb during gait
gait time percentage of left lower limb | after 3 months of treatment
  the time of stance and swing phases as a percentage for left lower limb during gait

SECONDARY OUTCOMES:
level of function through GMFCS | before and after 3 months of treatment
  changing the level of function by using the GMFCS

CONTACTS AND LOCATIONS:
Overall Officials: Nahla Mohamed, lecturer, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy,Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No